CLINICAL TRIAL: NCT00245544
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Explore the Safety and Preliminary Efficacy of Oral MK0759 in the Treatment of Postherpetic Neuralgia
Brief Title: Safety and Preliminary Efficacy of MK0759 in Postherpetic Neuralgia (PHN)(0759-004)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0759-004; MK0759-004; 2005_078
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0759

SUMMARY:
The purpose of this study is to test the safety and effect of MK0759 in relieving neuropathic pain as experienced by patients with postherpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85; diagnosis of postherpetic neuralgia with pain having persisted at least 6 months; dissatisfied with current regimen of pain control; able to complete study questionnaires, patient diary, and comply with daily study medication

Exclusion Criteria:

* Women of childbearing potential; history or evidence of a condition that, in the opinion of the investigator, may interfere with the study interpretation (e.g., diabetic neuropathy or fibromyalgia) or pose undue risk to undergo the course of medication required by the study (e.g., unstable heart disease, morbid obesity, kidney or liver disease).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity recorded by the patient each evening using an 11-point Likert scale (0=no pain to 10=pain as bad as you can imagine). | Duration of Treatment

SECONDARY OUTCOMES:
Safety; Patient Global Impression of Change assessed at the end of each treatment period. | Duration of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC